CLINICAL TRIAL: NCT03128957
Title: Correlating Brain Tissue Oxygen Tension (PbrO2) and Regional Cerebral Oximetry (rSO2) in Normal Human Brain Under the Conditions of Changing Ventilation Strategy
Brief Title: Correlating Brain Tissue Oxygen and Regional Cerebral Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paul Picton, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00105648
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Varying cerebral oxygenation with varying ventilation (Experimental): Compare oxygenation under conditions of varying ventilation strategy. Low end tidal CO2/Low inspired oxygen vs High end tidal CO2/high inspired oxygen
  Interventions: Device: IVOS cerebral oximeter; Device: Licox cerebral oxygenation monitor; Other: Cerebral oxygenation

INTERVENTIONS:
Device: IVOS cerebral oximeter — Measuring percutaneous cerebral oxygenation secondary to changing end tidal carbon dioxide and inspired oxygen fraction.
Device: Licox cerebral oxygenation monitor — Measuring tissue cerebral oxygenation secondary to changing end tidal carbon dioxide and inspired oxygen fraction.
Other: Cerebral oxygenation — Measuring cerebral oxygenation with varying ventilation strategy

SUMMARY:
Controversy surrounds the use of regional cerebral oximetry (rSO2) as a measure of true cerebral oxygenation because of extracranial signal contamination and unmeasured confounding of cerebral a:v ratio. The measurement of brain tissue oxygen (PbrO2) has been used in routine neurosurgery and has been shown to reliably demonstrate cerebral hypoxia following severe head injury. It is the most direct measure of cerebral oxygenation. Here, we test the hypothesis that there is a correlation between PbrO2 and rSO2 under conditions of varying inspired oxygen fraction and the varying partial pressure of carbon dioxide in arterial blood in uninjured, normal human brain.

Patients who are scheduled for elective removal of secondary cerebral metastases under general anesthesia will be recruited following written informed consent obtained by a study team member during their preoperative evaluation. BIS and rSO2 optodes will be applied, before induction of anesthesia, by a single researcher on both sides of the patient's forehead, as recommended by the manufacturer. General anesthesia will be maintained by total intravenous anesthesia (TIVA) with a combination of propofol (80-150 mcg/kg/min) and remifentanil (0.05-0.1 mcg/kg/min) targeted to a Bispectral Index range 40-60 (BIS; Covidien, Boulder, CO). Following craniotomy, the LICOX probe will be placed under direct vision into an area of normal brain within the tumor excision canal by the attending neurosurgeon. During a pause in surgery FIO2 and minute ventilation will be sequentially adjusted to achieve the following pairs of ventilation set points: 1) FIO2 0.3 and paCO2 30mmHg, 2) FIO2 1.0 and paCO2 40mmHg. After ≥5 minutes at each set point FIO2, PaCO2, rSO2 and PbrO2 will be recorded as a "snap-shot".

A sample size of 15 achieves an 80% power with a one-sided type I error of 5% to detect a positive correlation of 0.6 (from the null hypothesis of no correlation) between changes in PbrO2 and changes in rSO2 subsequent on alterations made in ventilation strategy. Correlation will be measured using Pearson's Correlation. P values < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective removal of secondary cerebral metastases under general anesthesia.

Exclusion Criteria:

* Patients will be excluded if they refuse to give consent, have evidence of elevated intracranial pressure on preoperative CT scan, have coagulopathy, are taking therapeutic agents known to increase bleeding risk, have a history of cardiovascular disease, cerebrovascular disease, suffer from respiratory failure, or are not fluent English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Picton, MB ChB, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 subjects were consented, two were excluded for logistical reasons prior to any data collection.
Period: Overall Study
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Regional Cerebral Oximetry (RSO2) and Cerebral Oxygen Tissue Tension (PbrO2).
Description: Correlation - correlation coefficient between cerebral oxygenation measured by Licox and INVOS oxygen measurement systems subsequent upon changes in ventilation strategy
  Spearman correlation describes the strength of the monotonic relationship between two measures and is bounded between -1 and 1. Negative values indicate an inverse relationship while positive values mean that the variables move in tandem.
  [Example of correlation coefficient in CT.gov: NCT02318667]
Time Frame: Time required for cerebral oxygenation to reach equilibrium following a change in ventilation - typically less than 20 minutes
Population: One subject's data was identified as an extreme value using the Tuckey Fences approach and was excluded from primary analysis.
Measure: Number; unit: Spearman Correlation (rs) Coefficient
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
Number analyzed (Participants) | 9
Spearman Correlation (rs) Coefficient | .5
Statistical Analysis 1: Comparison: Varying Cerebral Oxygenation With Varying Ventilation; Non-parametric covariance adjusted Spearman's correlation ρ_s. To test the Null that Ho: ρ_s.=0 vs alternative that Ha: ρ_s.≠0, we used a method that calculates the probability that it would be greater than or equal to the observed ρ ̂, given the null hypothesis, by using a permutation test. An advantage of this approach is that it automatically takes into account the number of tied data values in the sample and the way they are treated in computing the rank correlation; Test type: Equivalence — Given the small sample permutation are feasible; p = 0.036, permutation test; Given the non-parametric nature of spearman's correlation coefficient and a small sample we used a permutation test to calculate p-values

2. Secondary Outcome: Changes in PbrO2 Resultant Upon Changes in End Tidal Carbon Dioxide and Inspired Oxygen Fraction
Description: PbrO2 - measured in millimeters of mercury(mmHg); Steady State PbrO2 Upon Changes in End Tidal Carbon Dioxide and Inspired Oxygen Fraction after Equilibration for each Set Point
Time Frame: as for outcome 1
Population: One participant was identified as an extreme value using the Tuckey Fences approach and was excluded from final analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
Number analyzed (Participants) | 9
mmHg
  Set point 1 (FiO2 0.3 and PaCO2 30 mmHg) | 6.0 [4.0 to 11.3]
  Set point 2 (FiO2 1.0 and PaCO2 40 mmHg) | 22.5 [9.8 to 43.6]
Statistical Analysis 1: Comparison: Varying Cerebral Oxygenation With Varying Ventilation; Set point 1 (FiO2 0.3 and PaCO2 30 mmHg) compared to set point 2 (FiO2 1.0 and PaCO2 40 mmHg); Test type: Superiority; p = 0.015, Kruskal-Wallis

3. Secondary Outcome: Changes in rSO2 Resultant Upon Changes in End Tidal Carbon Dioxide and Inspired Oxygen Fraction
Description: rSO2 - %saturation; Steady State rSO2 Upon Changes in End Tidal Carbon Dioxide and Inspired Oxygen Fraction after Equilibration for each Set Point
Time Frame: as for outcome 1
Population: One subject was identified as an extreme value using the Tuckey Fences approach and was excluded from final analysis.
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
Number analyzed (Participants) | 9
percentage saturation
  Set Point 1 (FiO2 0.3 and PaCO2 30 mmHg) | 68.0 [62.5 to 80.5]
  Set Point 2 (FiO2 1.0 and PaCO2 40 mmHg) | 83.0 [74.0 to 90.0]
Statistical Analysis 1: Comparison: Varying Cerebral Oxygenation With Varying Ventilation; Set point 1 (FiO2 0.3 and PaCO2 30 mmHg) compared to set point 2 (FiO2 1.0 and PaCO2 40 mmHg); Test type: Superiority; p = 0.047, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Data were collected intraoperatively, and postoperatively for 24 hours.
Arm/Group | Varying Cerebral Oxygenation With Varying Ventilation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03128957/Prot_SAP_000.pdf